CLINICAL TRIAL: NCT05244733
Title: Culture and Well-Being for Latinos: Study Protocol for Cultural-Social Engagement and Suicide Among Hispanics (K23MH125078)
Brief Title: Culture and Well-Being for Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Caroline Silva, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006325; K23MH125078 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Social Isolation; Loneliness; Suicidal Ideation
MeSH Terms: conditions — Social Isolation; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Engage (S-ENGAGE) (Experimental): S-ENGAGE is a skills-based psychotherapy that focuses on helping patients engage in meaningful rewarding social activities. Subjects will receive 10 one-hour individual sessions of S-ENGAGE over 10 weeks.
  Interventions: Behavioral: Social Engage (S-ENGAGE)
- The Healthy Lifestyles Education Program (Placebo Comparator): The healthy lifestyles education program consists of a notebook containing evidence-based educational material on mental health, physical activity, and information on community resources. Study staff meet with participants once, individually, for 1 hour to review each section and answer questions participants might have.
  Interventions: Behavioral: The Healthy Lifestyles Education Program

INTERVENTIONS:
Behavioral: Social Engage (S-ENGAGE) — S-ENGAGE uses the process of action planning to foster sustained behavior change. Action planning involves: 1) select a goal; 2) develop ideas to meet this goal; 3) choose one or more of these ideas; 4) identify concrete steps to implement the goal (i.e., form an action plan); 5) identify and address barriers if needed.
  Arms: Social Engage (S-ENGAGE)
Behavioral: The Healthy Lifestyles Education Program — The healthy lifestyles education program is a self-guided psychoeducational program, including a notebook containing evidence-based educational material on mental health, physical activity, and information on community resources.
  Arms: The Healthy Lifestyles Education Program

SUMMARY:
The proposed K23 study is an intervention study using an experimental therapeutics approach. This pilot RCT asks: "Does SOCIAL-ENGAGE increase cultural-social engagement and decrease suicide risk among Spanish-speaking adults?" We will first optimize a behavioral intervention - SOCIAL ENGAGE (S-ENGAGE) - for target engagement using human-centered design approaches with Spanish-speaking adults at risk for suicide (n=5) and then conduct a pilot RCT (n=60) to test target engagement (cultural-social engagement) and clinical impact (suicide risk) of S-ENGAGE with this population. The ultimate goal is for S-ENGAGE to be offered as a suicide prevention program for Hispanics at risk for suicide.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Hispanic/Latino adult (age 18+);
* Primary Spanish-Speaker;
* Patient in the UR health system;
* Low cultural-social engagement (i.e., score ≤ 2 on the adapted Berkman-Syme Social Network Index);
* Elevated suicide risk (i.e., presence of passive or active suicide ideation in the past month on the Columbia-Suicide Severity Rating Scale [C-SSRS]).

Exclusion Criteria:

* Medical or psychiatric comorbidities that impair ability to consent (e.g., active psychotic or manic episode, cognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Change in Cultural-Social Engagement (A) | Baseline and 10 weeks
  Average number of cultural-social interactions (measured via EMA), with greater number indicating greater cultural-social engagement (i.e., better outcome).
Change in Cultural-Social Engagement (B) | Baseline and 10 weeks
  Time spent in positive Spanish-language conversations (measured via passive monitoring of conversations), with more time indicating greater cultural-social engagement (i.e., better outcome).
Change in Cultural-Social Engagement (C) | Baseline and 10 weeks
  Number of visits to cultural-social settings outside the home (measured via GPS), with greater number indicating greater cultural-social engagement (i.e., better outcome).
Change in Cultural-Social Engagement (D) | Baseline and 10 weeks
  Self-reported feelings of belonging to Hispanic cultural groups (measured via EMA with the Interpersonal Needs Questionnaire), with greater scores indicating greater cultural-social engagement (i.e., better outcome).

SECONDARY OUTCOMES:
Change in Suicide Risk (A) | Baseline and 10 weeks
  Reasons for living total score, measured by the Reasons for Living Inventory, with 48 items rated from 1 to 6, with greater scores indicating greater importance for reasons for living (i.e., better outcome).
Change in Suicide Risk (B) | Baseline and 10 weeks
  Suicide ideation total score, measured by the Beck Scale for Suicide Ideation, with scores ranging from 0 to 38, with greater scores indicating greater suicide ideation (i.e., worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No